CLINICAL TRIAL: NCT04201808
Title: Efficacy and Safety of Tenofovir Alafenamide in Chronic Hepatitis B Patients With Suboptimal Response Following Nucleos(t)Ide Therapy
Brief Title: Efficacy and Safety of TAF in Patients With Suboptimal Response to Other Nucleos(t)Ides
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New Discovery LLC (Industry)
Collaborators: Beijing Ditan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-CN-320-5556
Record Dates: First submitted 2019-12-06; First posted 2019-12-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: This is single-arm, multicenter cohort study evaluating the efficacy, safety, and tolerability of TAF monotherapy in Asian CHB adults with SOR to the nucleos(t)ide therapy by assessing the HBV DNA suppression over a duration of 48 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Intervention Group (Experimental): All approximately 100 patients experienced previous suboptimal response to other direct acting antivirals. Patients must have received nucleos(t)ide therapy consisting of LAM/LdT/ADV and its combinations with other second-line antivirals for 24 weeks, or with the first-line antiviral ETV or any antiviral combinations containing ETV for 48 weeks with medication adherence. All patients in this study are in the same arm.
  Interventions: Drug: Tenofovir Alafenamide 25 MG

INTERVENTIONS:
Drug: Tenofovir Alafenamide 25 MG — All patients will receive Tenofovir Alafenamide, 25mg PO, to treat chronic hepatitis B and their previous suboptimal response over the study duration of 48 weeks. Patients will be followed every 12 weeks for medication adherence, medication refill, and follow up as per standard of care.
  Other Names: Vemlidy

SUMMARY:
Both tenofovir disoproxil fumarate (TDF) and tenofovir alafenamide (TAF) are potent antiviral agents for hepatitis B virus (HBV) and recommended by the American Association for the Study of Liver Disease (AASLD) as well as the European Association for the Study of Liver (EASL) guidelines for the treatment of nucleos(t)ide therapy induced HBV resistance. However, it is not clear if chronic hepatitis B (CHB) patients with nucleos(t)ide treatment experience without genotypic mutations would be benefit from TAF therapy. Previous studies have observed that suboptimal response (SOR) following antiviral therapy with nucleos(t)ide treatment is associated with an increased risk of subsequent treatment failure and viral resistance. It remains unclear whether switching to TAF is a reasonable approach in patients with SOR to second-line antivirals Lamivudine (LAM)/ Telbivudine (LdT)/ Adefovir Dipivoxil (ADV) and its combinations with other second-line antivirals for 24 weeks, or SOR to the first-line antiviral Entecavir (ETV) or any antiviral combinations containing ETV for 48 weeks. This study is aimed to determine how the aforementioned patients with SOR to nucleos(t)ide treatment respond to TAF monotherapy. The investigator's study will provide evidence base for therapy selection in SOR patients, especially in China where the majority of patients with CHB are treated with nucleos(t)ide therapy.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter cohort study evaluating the efficacy, safety, and tolerability of TAF monotherapy in in Asian CHB adults with SOR to the nucleos(t)ide therapy by assessing the HBV DNA suppression in 48 weeks. Approximately one hundred adults who received the aforementioned nucleos(t)ide therapy will be prospectively enrolled during the period from December 2019 to June 2021. Subjects will be enrolled by medical clinic in about 10 university centers in different regions in China. Approximately 10-15 consecutive eligible patients will be enrolled from each participating sites. This study will be conducted in accordance with the guidelines of Good Clinical Practices (GCPs) including Institutional Review Board (IRB) approval and consent will be applied. Patient identification (ID) will be de-identified for submitting to the central database for analyses from all study sites. Free TAF treatment will be provided to all enrolled patients for 48 weeks. Patients will be under the local standard of care upon the completion of the current study.

Patients aged 18-80 with CHB infection who had received nucleos(t)ide therapy over 24 weeks of LAM/LdT/ADV or 48 weeks of ETV with medication adherence, but failure to achieve the levels of HBV-DNA below 300 IU/mL will be eligible. Subjects will be excluded if they meet the following criteria: co-infected with HIV or other viral hepatitis; the serum levels of HBV DNA are too low (i.e. about 300 IU/mL) to be analyzed for the genotypic mutation(s); nucleos(t)ide resistant mutants have been detected at screening visit, patient is under a clinical research protocol of phase I-III development; unable to consent or unlikely to complete one year follow up after the enrollment; and other medical condition may affect the ability to participate the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18-80 years of age.
* Patients must have documented compensated and stable chronic hepatitis B defined by all of the following:

  * HBsAg persistently positive > 6 months.
  * Clinical history, physical findings, and test results are compatible with compensated chronic hepatitis B
* Patients must have received nucleos(t)ide therapy consisting of LAM/LdT/ADV and its combinations with other second-line antivirals for 24 weeks, or with the first-line antiviral ETV or any antiviral combinations containing ETV for 48 weeks with medication adherence.
* Although having undergone therapy, patients have had failure to achieve the levels of HBV-DNA below 300 IU/mL.
* Patient is willing and able to comply with the study drug regimen and all other study requirements.
* Patient must understand the risk, and be willing and able to provide written informed consent to participate in the study.

Exclusion Criteria:

* Pregnant women, and women who are breastfeeding or who believe they may wish to become pregnant during the course of the study.
* Males and females of reproductive potential who are not willing to use an effective method of contraception during the study. For males, condoms should be used and for females, a barrier contraception method should be used in combination with one other form of contraception.
* Unwilling and/or unable to provide written informed consent
* Patients with CHB but are also co-infected with HIV or other viral hepatitis
* Patients whose serum levels of HBV DNA are too low (i.e. about 300 IU/mL) to be analyzed for the genotypic mutation(s) at the onset of this trial, i.e. baseline
* At the screening visit, nucleos(t)ide resistant mutants have been detected in the strain of HBV of the patient
* The patient is under a clinical research protocol of phase I-III development; unable to consent or unlikely to complete one year follow up after the enrollment; and other medical condition may affect the ability to participate the study.
* Decompensated liver disease defined as direct (conjugated) bilirubin ≥ 1.2 Upper Limit of Normal (ULN); Prothrombin Time (PT) ≥ 1.2 ULN, platelets ≤ 150,000/mm3, or serum albumin ≤ 3.5 g/dL
* Prior history of clinical hepatic decompensation (e.g., ascites, jaundice, encephalopathy) or variceal hemorrhage
* Serum α-fetoprotein ≥ 50 ng/mL
* Evidence of hepatocellular carcinoma (HCC)
* History of significant renal disease (e.g., nephrotic syndrome, renal dysgenesis, polycystic kidney disease, congenital nephrosis, acute tubular necrosis, other renal disease)
* History of significant bone disease (e.g., osteomalacia, chronic osteomyelitis, osteogenesis imperfecta, osteochondrosis, multiple bone fractures)
* Significant cardiovascular, pulmonary or neurological disease
* Evidence of a gastrointestinal malabsorption syndrome that may interfere with absorption of orally administered medications
* History of solid organ or bone marrow transplantation
* Ongoing therapy with any of the following: Nephrotoxic agents

  * Parenteral aminoglycoside antibiotics (e.g., gentamicin, tobramycin, amikacin)
  * Cidofovir
  * Cisplatin
  * Foscarnet
  * IV amphotericin B
  * IV pentamidine
  * Oral or IV ganciclovir
  * Cyclosporine
  * Tacrolimus
  * IV vancomycin
  * Chronic daily non-steroidal anti-inflammatory drug therapy
  * Competitors of renal excretion (e.g., probenecid) Systemic chemotherapeutic agents
  * Systemic corticosteroids
  * Interleukin-2 (IL-2) and other immunomodulating agents
* Investigational agents (except with the expressed approval of the lead investigators)

Note: administration of any of the above medications must be discontinued at least 30 days prior to the Baseline Visit and for the duration of the study period.

* Known hypersensitivity to the study drugs, the metabolites or formulation excipients
* Any other condition (including alcohol or substance abuse) or prior therapy that, in the opinion of the Investigators, would make the subject unsuitable for the study or unable to comply with dosing requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
this study seeks to evaluate the efficacy of TAF in Asian CHB adults with a proven SOR to previous nucleo(t)side therapy by assessing the percentage of patients who achieve HBV DNA viral suppression over a time span of 48 weeks. | 48 weeks
  In this study, HBV DNA viral suppression is defined as a HBV DNA level <20 IU/mL, and previous nucleo(t)side therapy is defined as treatments including LAM, LdT, ADV, and ETV before switching to TAF. The parameters for SOR will be set as patients who exhibit a 1 log10 IU/mL decrease in HBV DNA with medication adherence, but still present with an HBV DNA level of >300 IU/mL and has no detectable genotype mutation(s) when treated with the second-line antivirals LAM/LdT/ADV and its combinations with other second-line antivirals for 24 weeks, or treated with the first-line antiviral ETV or any antiviral combinations containing ETV for 48 weeks.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events in Patients as stratified by the CTCAE v 5.0 | At 12, 24, 36, and 48 weeks
  Assess the percentage of Asian CHB adults with SOR to nucleos(t)ide therapy who have adverse events during the study, graded by the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Percentage of Patients Who Discontinue the Therapy Due to Issues with Tolerability | At 12, 24, 36, and 48 weeks
  To evaluate the frequency of treatment discontinuation in patients who can not tolerate TAF therapy
Percentage of patients with Alanine transferase (ALT) levels within the normal limit | 48 weeks
  To calculate the percentage of patients at the end of 48 weeks whose ALT (U/L) levels stay within the normal limit in response to TAF therapy in Asian adults with CHB infection who are SOR to nucleos(t)ide therapy.
Percentage of patients with Aspartamine transferase (AST) levels within the normal limit | 48 weeks
  To calculate the percentage of patients at the end of 48 weeks whose AST (U/L) levels stay within the normal limit in response to TAF therapy in Asian adults with CHB infection who are SOR to nucleos(t)ide therapy.
Percentage of patients who experience loss/seroconversion of HBsAg and/or HBeAg during the study. | 48 weeks
  Assess the percentage of patients who loss/seroconversion of HBsAg or/and HBeAg during the study. Loss is defined by a test showing a negative HBsAg/HBeAg result at the end of the trial, given a positive respective test result at baseline. A seroconversion is defined as a test showing a negative HBsAg and a positive HBsAb result, or a negative HBeAg and a positive HBeAb result at the end of the trial, given a positive HBsAg/HBeAg test result at baseline.
Percentage of patients with detectable drug resistance mutations | 48 weeks
  To evaluate the incidence of drug resistance and drug resistance mutations in 48 weeks of TAF treatment if patients have HBV DNA levels >300 IU/mL. Drug resistance by population sequencing and genotyping will be done for these patients.
Percentage of patients who have skipped TAF treatment during the study | 48 weeks.
  Assess the medication compliance on patients and compare the two sub-groups of patients who will be stratified by the levels of HBV DNA using the cut of of 20 IU/mL at 48 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Q Pan, MD, Principal Investigator — NYU Langone Health; Wen Xie, MD, Study Director — Capital Medical University
Locations (10):
- China (10):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Liver Research Center, The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Wuhan Union Hospital, Tongji Medical College (TJMC), Huazhong University of Science and Technology (HUST), Wuhan, Hubei
  - Shengjing Hospital of China Medical University, Shengyang, Liaoning
  - Department of Infectious Diseases, Xi'an Jiaotong University Second Affiliated Hospital, Xi'an, Shaanxi
  - Huashan Hospital Fudan University, Jing’an, Shanghai Municipality
  - The Third Hospital of Hebei Medical University, Hebei, Shijiazhuang

REFERENCES:
- [Background] Agarwal K, Brunetto M, Seto WK, Lim YS, Fung S, Marcellin P, Ahn SH, Izumi N, Chuang WL, Bae H, Sharma M, Janssen HLA, Pan CQ, Celen MK, Furusyo N, Shalimar D, Yoon KT, Trinh H, Flaherty JF, Gaggar A, Lau AH, Cathcart AL, Lin L, Bhardwaj N, Suri V, Mani Subramanian G, Gane EJ, Buti M, Chan HLY; GS-US-320-0110; GS-US-320-0108 Investigators. 96 weeks treatment of tenofovir alafenamide vs. tenofovir disoproxil fumarate for hepatitis B virus infection. J Hepatol. 2018 Apr;68(4):672-681. doi: 10.1016/j.jhep.2017.11.039. Epub 2018 Jan 17. PMID 29756595
- [Background] Buti M, Gane E, Seto WK, Chan HL, Chuang WL, Stepanova T, Hui AJ, Lim YS, Mehta R, Janssen HL, Acharya SK, Flaherty JF, Massetto B, Cathcart AL, Kim K, Gaggar A, Subramanian GM, McHutchison JG, Pan CQ, Brunetto M, Izumi N, Marcellin P; GS-US-320-0108 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of patients with HBeAg-negative chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):196-206. doi: 10.1016/S2468-1253(16)30107-8. Epub 2016 Sep 22. PMID 28404092
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Lu L, Yip B, Trinh H, Pan CQ, Han SH, Wong CC, Li J, Chan S, Krishnan G, Wong CC, Nguyen MH. Tenofovir-based alternate therapies for chronic hepatitis B patients with partial virological response to entecavir. J Viral Hepat. 2015 Aug;22(8):675-81. doi: 10.1111/jvh.12368. Epub 2014 Nov 24. PMID 25417914
- [Background] Pan CQ, Chan S, Trinh H, Yao A, Bae H, Lou L. Similar efficacy and safety of tenofovir in Asians and non-Asians with chronic hepatitis B. World J Gastroenterol. 2015 May 14;21(18):5524-31. doi: 10.3748/wjg.v21.i18.5524. PMID 25987775
- [Background] Pan CQ, Hu KQ, Yu AS, Chen W, Bunchorntavakul C, Reddy KR. Response to tenofovir monotherapy in chronic hepatitis B patients with prior suboptimal response to entecavir. J Viral Hepat. 2012 Mar;19(3):213-9. doi: 10.1111/j.1365-2893.2011.01533.x. Epub 2011 Oct 17. PMID 22329376
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] Tong MJ, Pan CQ, Han SB, Lu DS, Raman S, Hu KQ, Lim JK, Hann HW, Min AD. An expert consensus for the management of chronic hepatitis B in Asian Americans. Aliment Pharmacol Ther. 2018 Apr;47(8):1181-1200. doi: 10.1111/apt.14577. Epub 2018 Feb 26. PMID 29479728